CLINICAL TRIAL: NCT00315276
Title: A 9-week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Finding Study to Evaluate the Efficacy and Safety of Modafinil as Treatment for Adults With Attention Deficit/Hyperactivity Disorder
Brief Title: Dose-Finding Study to Evaluate the Efficacy and Safety of Modafinil as Treatment for Adults With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1538/2027/AD/US
Record Dates: First submitted 2006-04-17; First posted 2006-04-18 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2007-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of modafinil administered once daily for 9 weeks at doses of 255, 340, 425, and 510 mg as treatment for adults with ADHD.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether modafinil at 255, 340, 425, or 510 mg'day is more effective than a placebo in alleviating the symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults as determined by the change from baseline in the total score from the investigator-completed Adult ADHD Investigator Symptoms Rating Scale (AISRS) the at endpoint (last post-baseline observation [week 9 or early termination]).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The patient is 18 to 65 years of age (inclusive) at the screening visit and is English speaking.
* At screening (after washout, if required) the patient meets the full Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for ADHD (combined type, predominantly inattentive subtype, or predominantly hyperactivity-impulsive subtype), for which symptoms were present for the age of 7 and symptoms have been persistent for at least the last 6 months, according to a psychiatric/clinical evaluation using the adult ADHD Clinical Diagnosis Scale, Version 1.2 (ACDS).
* The patient has a Hamilton Anxiety Scale (HAM-A) and a Hamilton Depression Scale (HAM-D) score less than 15.
* The patient has an AISRS total score of greater than 24 at the screening and baseline visits, and the difference in the total score from the screening visit to the baseline visit is less than 25%.
* The patient has a Clinical Global Impression of Severity of Illness (CGI-S) rating for ADHD of at least 4 at the baseline visit.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study. Acceptable methods of contraception include barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method, or intrauterine device [IUD].
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* The patient has a history or current diagnosis of schizophrenia, bipolar or other psychotic disorders, or clinical assessment of suicide risk.
* The patient has any current psychiatric comorbidity, including but not limited to depression or other mood disorder or anxiety disorder, that requires pharmacotherapy. Comorbidities will be assessed using selected modules (ie, psychosis, substance abuse, mood disorder, anxiety disorders) of the Structured Clinical Interview for DSM-IV-TR (SCID).
* The patient has a current diagnosis of a clinically significant sleep disorder.
* The patient is intellectually challenged, as determined by the investigator.
* The patient is satisfied with current ADHD medication and has no unacceptable medication side effects.
* The patient has previously used modafinil.
* The patient is using other prescription medications for ADHD with psychoactive properties (eg, amphetamine, dextroamphetamine, methylphenidate, pemoline, atomoxetine) at the baseline visit.
* The patient has had drug or alcohol abuse or dependence within the last 6 months.
* The patient has used monoamine oxidase (MAO) inhibitors or selective serotonin reuptake inhibitors (SSRIs) within 2 weeks before the baseline visit.
* The patient has used an investigational drug within 1 month before the baseline visit.
* The patient is pregnant or lactating. (Any patients becoming pregnant during the study will be withdrawn from the study).
* The patient has any clinically significant uncontrolled medical conditions (treated or untreated).
* The patient has a clinically significant deviation from normal in the physical examination.
* The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2006-05; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Neurology Clinical Study Centers, LLC, Little Rock, Arkansas
  - Bay Area Research Institute, Lafayette, California
  - Pharmacology Research Institute, Northridge, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - UCSD Medical Center, San Diego, California
  - Clinical Neuroscience Solution, Inc., Orlando, Florida
  - University of Illinois, Chicago, Illinois
  - Michael J. Reiser, MD, LLC, Lexington, Kentucky
  - Adult ADD Center of Maryland, Lutherville, Maryland
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester, Michigan
  - CRI WorldWide, LLC, Clementon, New Jersey
  - New York University, New York, New York
  - Summit Research Network Inc., Portland, Oregon
  - CRI WorldWide, LLC, Philadelphia, Pennsylvania
  - South East Health Consultants, LLC, Charleston, South Carolina
  - Clinical Neuroscience Solution, Memphis, Tennessee
  - Neuropsychiatric Associates, Woodstock, Vermont